CLINICAL TRIAL: NCT06747702
Title: Effect of Integrated Workouts on Injury Prevention in Overhead Athletes
Brief Title: Injury Prevention Programs in Overhead Athletes
Acronym: IPOverhead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Responsible Party: Principal Investigator, Monica Solana Tramunt, PhD, University Ramon Llull
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Injury prevention Overhead
Record Dates: First submitted 2024-12-06; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Shoulder Impingement Syndrome; Shoulder Injury; Shoulder Pain Chronic; Shoulder Joint Limitation; Shoulder Flexibility
Keywords: Injury prevention; Glenohumeral rotation deficits; Overhead athletes; shoulder pain; Shoulder instability; Shoulder mobility; Shoulder exercises; Shoulder symetries; Shoulder Asymetries; Shoulder stability; Shoulder strength; Escapulahumeral complex
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware of whether they belong to the experimental or control group. They will receive instructions on their workout regimen without information on the study's hypothesis regarding functional prevention training.
  Individuals conducting pre- and post-intervention assessments (e.g., EMG analysis, ROM measurements, proprioception tests) will not be informed of the participant group allocation. This prevents bias in data collection and interpretation.
  Data will be anonymized before analysis, and analysts will not have access to group identifiers during the statistical evaluation phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group: Participants in this group will undergo the intervention (Experimental): Participants for the injury prevention program
  Interventions: Other: Injury prevention workout
- Control group (No Intervention): Participant with same training program that will not be involved in the intervention although they will follow same specific sport practice

INTERVENTIONS:
Other: Injury prevention workout — The injury prevention workout consisted on engaging on a prevention program from 1 day to 8 weeks where the participants will develop functional sport exercises to prevent shoulder injuries or pain in overhead sports.
  Arms: Experimental Group: Participants in this group will undergo the intervention

SUMMARY:
To evaluate and describe the effect of performing an integrated injury prevention exercises on the variables considered as injury risk factors in overhead athletes

DETAILED DESCRIPTION:
To evaluate and describe the effect of performing fast or 6-8 weeks injury prevention programs on the variables considered as injury risk factors in overhead athletes as glenohumeral rotational range of motion or muscle activation pattern and asymmetries.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent according last version ogf Helsinky Declaration.
* Be involved in a overhead sport for a minimum of 2 years.

Exclusion Criteria:

* Have some pain or disconfort to develop the outcome measurements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Shoulder ROM | From enrollment to the end of the intervention at 8 weeks. Follow-up at 12-weeks
  Shoulder rotational range of movement will be measured made by a single experienced examiner with the IMU Output Capture (Output V2 Unit, Ireland). The IMU will be calibrated prior to ROM testing according to the device instructions. The IMU will be securely attached to the participant's forearm with a self-adhering strap, 10 cm distal to the lateral epicondyle. Measurements will be sent wirelessly to a tablet and subsequently transferred to the Output Hub specific software to calculate ROM
Muscle RMS | From enrollment to the end of the intervention at 8 weeks. Follow-up at 12-weeks
  Escapular complex muscular activation EMG recording will be measured with the mDurance® device (mDurance® Solutions SL, Granada, Spain). The mDurance® system consisted of an EMG Shimmer3 unit (Realtime TechnologiesLtD, Dublin, Ireland). Muscles-activity data were obtained using a validated surface electromyography (EMG) system. This novel system includes a us-er-friendly software, and a light hardware, which make it more affordable and accessible for clinicians and sport trainers. The mDurance® system consisted of an EMG Shimmer3 unit (Realtime TechnologiesLtD, Dublin, Ireland). The unit has a bipolar surface elec-tromyography bipolar sensor for the acquisition of muscle activity. Each Shimmer3 has two channels, with a sampling rate of 1024 Hz applying a bandwidth of 8.4 Hz, and a 24-bit signal with an overall amplification of 100 to10,000 v/v [41]. This device is valid and reliable for recording muscle activity during a functional task (ICC = 0.916; 95% CI = 0.831-0.958)
Muscles Asymetries | From enrollment to the end of the intervention at 8 weeks. Follow-up at 12-weeks
  Diferences in % the muscle activation of the interescapular muscle complex by EMG. These recording will be also performed with the mDurance® device (mDurance® Solutions SL, Granada, Spain). The mDurance® system consisted of an EMG Shimmer3 unit (Realtime TechnologiesLtD, Dublin, Ireland) . This device is valid and reliable for recording muscle activity during a functional task (ICC = 0.916
Shoulder proprioception | From enrollment to the end of the intervention at 8 weeks. Follow-up at 12-weeks
  The Ability of recognizing a specific glenohumeral rotational range of movement degrees we will use the IMU Output Capture (Output V2 Unit, Ireland). The IMU was calibrated prior to ROM testing according to the device instructions. The IMU was securely attached to the participant's forearm with a self-adhering strap, 10 cm distal to the lateral epicondyle. Measurements were sent wirelessly to a tablet and subsequently transferred to the Output Hub specific software to calculate ROM

CONTACTS AND LOCATIONS:
Locations (1):
- FPCEE Blanquerna, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Not proceed

REFERENCES:
- [Background] McKenzie A, Larequi SA, Hams A, Headrick J, Whiteley R, Duhig S. Shoulder pain and injury risk factors in competitive swimmers: A systematic review. Scand J Med Sci Sports. 2023 Dec;33(12):2396-2412. doi: 10.1111/sms.14454. Epub 2023 Jul 28. PMID 37515375
- [Background] Cools AM, Johansson FR, Borms D, Maenhout A. Prevention of shoulder injuries in overhead athletes: a science-based approach. Braz J Phys Ther. 2015 Sep-Oct;19(5):331-9. doi: 10.1590/bjpt-rbf.2014.0109. Epub 2015 Sep 1. PMID 26537804
- [Background] Wright AA, Ness BM, Donaldson M, Hegedus EJ, Salamh P, Cleland JA. Effectiveness of shoulder injury prevention programs in an overhead athletic population: A systematic review. Phys Ther Sport. 2021 Nov;52:189-193. doi: 10.1016/j.ptsp.2021.09.004. Epub 2021 Sep 14. PMID 34560586
- [Background] Liaghat B, Pedersen JR, Husted RS, Pedersen LL, Thorborg K, Juhl CB. Diagnosis, prevention and treatment of common shoulder injuries in sport: grading the evidence - a statement paper commissioned by the Danish Society of Sports Physical Therapy (DSSF). Br J Sports Med. 2023 Apr;57(7):408-416. doi: 10.1136/bjsports-2022-105674. Epub 2022 Oct 19. PMID 36261251
- [Background] Schwank A, Blazey P, Asker M, Moller M, Hagglund M, Gard S, Skazalski C, Haugsbo Andersson S, Horsley I, Whiteley R, Cools AM, Bizzini M, Ardern CL. 2022 Bern Consensus Statement on Shoulder Injury Prevention, Rehabilitation, and Return to Sport for Athletes at All Participation Levels. J Orthop Sports Phys Ther. 2022 Jan;52(1):11-28. doi: 10.2519/jospt.2022.10952. PMID 34972489
- [Background] Cools AM, Maenhout AG, Vanderstukken F, Decleve P, Johansson FR, Borms D. The challenge of the sporting shoulder: From injury prevention through sport-specific rehabilitation toward return to play. Ann Phys Rehabil Med. 2021 Jul;64(4):101384. doi: 10.1016/j.rehab.2020.03.009. Epub 2020 Apr 29. PMID 32320753
- [Derived] Solana-Tramunt M, Bofill-Rodenas A. Motor imagery enhances core training effects on lumbar proprioception in elite swimmers: a randomized controlled trial. Front Physiol. 2025 Sep 1;16:1667536. doi: 10.3389/fphys.2025.1667536. eCollection 2025. PMID 40959125